CLINICAL TRIAL: NCT06411782
Title: Investigation of the Effect of the Foam Roller Method Applied to the Sternocleidomastoid Muscle After Respiratory Muscle Fatigue
Brief Title: The Effect of Foam Roller Applied to the SCM Muscle on Respiratory Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foam Roller on SCM Muscle
Record Dates: First submitted 2024-05-04; First posted 2024-05-13 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Adults; Inspiratory Muscle Training
Keywords: Foam Roller; Sternocleidomastoid Muscle; Inspiratory Muscle Training; MIP

STUDY DESIGN:
Intervention Model Description: The study is a cross-controlled study. Inspiratory muscle training (IMT) training will be performed on the subjects, and then FR will be applied to the Right SCM muscle. A 1 week purification period will be given. Later, after the IMT study, FR will be applied to the Left SCM muscle. All evaluation parameters will be repeated before and after the applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam Roller Group (Experimental): Inspiratory muscle training will be done with a resistive exercise device at 80% of MIP max and for 30 breaths. After training, foam roller application will be applied to the right sternocloideomastoid muscle.
  Interventions: Device: Foam roller; Device: Inspiratory muscle training
- Non Foam Roller Group (Experimental): Inspiratory muscle training will be done with a resistive exercise device at 80% of MIP max and for 30 breaths. Foam roller application will not be done.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Foam roller — In foam roller application, a partitioned FR from the Trigger Point Grid 2.0 brand, measuring 33x14 cm and weighing 0.9 kg, with an inner part made of polyvinylchloride (PVC), will be used. Participants will roll the segmented FR with slight flexion-extension by placing the FR on the SCM muscle to apply FR from the starting point to the end point of that muscle region for the selected SCM muscle, with the person in the side stance position against the wall. This action will consist of 3 sets of 1 minute each, with a 30-second rest period between each set. It will be applied once for each region, including the right and left SCM muscle.
  Arms: Foam Roller Group
Device: Inspiratory muscle training — Inspiratory muscle training will be done with a resistive exercise device at 80% of MIP max and for 30 breaths.

SUMMARY:
The aim of this study is to examine the acute effect of the foam roller (FR) method applied to the sternocleidomastoid (SCM) muscle after respiratory muscle fatigue on joint range of motion (ROM), accessory respiratory muscle activity and muscle strength.

The aim of this study is to examine the changes in fatigue and pain symptoms by applying relaxation on the tense fascia and shortened muscle as a result of resistance training, and the effect of these changes in the sternocleidomastoid (SCM) muscle on joint range of motion (ROM) and muscle strength in healthy male or female participants aged 18-30.

In line with the investigators' results, it may be recommended to add foam roller (FR) to the accessory respiratory muscles in the pulmonary rehabilitation program in patients with chronic lung diseases. For this reason, the investigators think that it will provide clinical and scientific benefits.

The investigators believe that it will lead studies to add foam roller (FR) to the pulmonary rehabilitation program in patients with chronic lung diseases. Participants will be informed about the risks and benefits of participating in the study and a voluntary consent form will be signed. Participants will be given a demographic data form before starting the study and will be asked to fill it out. The hypermobility value will be measured according to the Beighton score before the participants start the tests. After the inspiratory muscle training (IMT) study, foam roller (FR) will be applied to the right sternocleidomastoid (SCM) muscle. A one week washout period will be given. Afterwards, the cases will be applied foam roller (FR) to the left sternocleidomastoid (SCM) muscle after the inspiratory muscle training (IMT) study. All evaluation parameters will be repeated before and after the applications. Maximum inspiratory pressure measurement, range of motion (ROM) measurements, muscle strength tests, flexibility with a myotony measuring device, electromyography (EMG) measurements will be made before the study one by one.

DETAILED DESCRIPTION:
The sternocleidomastoid muscle (SCM) is one of the largest cervical muscles located in the superficial layer of the neck region. The primary movements of the muscle are rotation and lateral flexion. Sternocleidomastoid (SCM) tends to be overactive in many people. In general, when abnormal postures and abnormal positions are adopted, they have to work harder to help stabilize the neck area and thus the head. It is also the auxiliary respiratory muscle for breathing along with the scalene muscles. For this reason, it has been reported in the literature that in patients with chronic lung diseases who have low respiratory capacity, tension and trigger points in the sternocleidomastoid (SCM) occur due to overwork of this muscle all day.

Foam Roller (FR) application is generally used to create pressure on soft tissues by using body weight and relaxation is achieved in the muscle. The aim of our study is to examine the acute effect of the foam roller (FR) method applied to the sternocleidomastoid (SCM) muscle after inspiratory muscle training (IMT) on range of motion (ROM) and muscle strength in healthy young adults. When the studies in the literature were examined, it was concluded that there was no study examining the effect of foam roller (FR) on sternocleidomastoid (SCM) before. In addition, there is no study examining the use of foam roller (FR) after inspiratory muscle training.

First of all, the target group (healthy adults) determined for the project will be participants, taking into account the inclusion and exclusion criteria. Each participant will sign the Voluntary Consent Form and participate in the study. Participants will be asked to fill out a demographic data form before starting the study and hypermobility values will be measured according to the Beighton score before starting the tests. Sternocleidomastoid (SCM) is an accessory respiratory muscle located in the neck. Due to the sensitivity of its location and function, it is important to perform the foam roller (FR) application with the right technique. For this reason, all volunteers participating in the investigators' study will be informed about the anatomical structure and kinesiological nature of the sternocleidomastoid (SCM) muscle and the foam roller (FR) application will be taught. After the selection and informing of the volunteers, the cases before the study one by one; measurement of maximum inspiratory pressure (MIP), range of motion (ROM) measurements, muscle activity measurement with electromyography (EMG), muscle strength tests, flexibility status parameters will be measured with a myotony measuring device. After all evaluations have been made, 30 breaths will be applied with 2 repetitions of inspiratory muscle training (IMT) with a Power Breathe device, 80% of the Maximum Inspiratory Pressure (MIP). After inspiratory muscle training (IMT), foam roller (FR) application on the sternocleidomastoid (SCM) muscle will be applied with 3 sets of 1 minute and a 30-second listening period between each set. 27 healthy cases will be included in our study. After the inspiratory muscle training (IMT) study, first foam roller (FR) will be applied to the right sternocleidomastoid (SCM) muscle in each included case, and then it will be evaluated with the evaluation criteria. After a 1 week washout period, foam roller (FR) will be applied to the left sternocleidomastoid (SCM) muscle after inspiratory muscle training (IMT) application. All measurements will be repeated immediately after the application and 15 minutes later.

The analysis of the data to be obtained will be carried out using the Statistical Package for the Social Sciences (SPSS) 25 package program.

As a result of the success of the project, it is thought that it will be a source of inspiration for new studies in patients with chronic lung diseases.

The project is an undergraduate thesis and if it is realized, it will contribute to the training of qualified and young researchers in our country.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults
* Not exercising regularly for the last 6 months
* To have participated in the study voluntarily
* Individuals without widespread visceral or musculoskeletal pain were included.

Exclusion Criteria:

* Using pain medication
* Soft tissue, muscle and bone injury
* Spinal cord or upper extremity injuries
* Fibromyalgia
* Cases treated with myofascial release
* Individuals who did not have hypermobility according to the Beighton score were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Muscle Stiffness and Muscle Tone of sternocleidomastoid muscle | 1 Hour
  Elasticity measurement will be evaluated with the MyotonPro brand device. Measurements will be made while the subjects are in the sitting position. Primarily, marking will be made between the adhesion site of the sternocleidomastoid (SCM) to the anterior surface of the manubrium sterni and the adhesion on the mastoid process of the temporal bone. Then the measurement will be made. The probe of the device (3 mm diameter) will be placed perpendicular to the skin surface with a constant preload (0.18 N).
Electromyographic activity level measurement of sternocleidomastoid muscle | During the intervention
  Trigno Avanti brand surface electromyography (EMG) measurement sensors will be used to record the superficial EMG signals. The skin area will be cleaned with alcohol. Contraction of the sternocleidomastoid (SCM) muscle will be achieved by performing SCM neck flexion movement and electrode placement will be determined by palpating the muscle midpoint. During the initial evaluation, after the inspiratory muscle training (IMT) study and after the foam roller (FR) application, measurements will be made from both SCM muscles.

SECONDARY OUTCOMES:
Sternocleidomastoid Muscle Strength Measurements | 1 Hour
  Lafayette hand dynamometer will be used. The device can give data such as peak power, time to reach peak power, total test time and average force in lbs. When the cervical region is in the neutral position, the device will be placed on the sternocleidomastoid muscle 90 degrees perpendicular and the make test protocol will be applied. Make test is the protocol of applying maximum force against the device by the person being measured while holding the dynamometer steady. Patients will be asked to perform lateral flexion, flexion and rotation movements in the supine position. And resistance will be applied in the opposite direction. Performing three repetitions will save the higher value. Measurements will be measured from the same part of the muscle each time, and the practitioner and the extremity performing the test will be the same.
Cervical joint range of motion | 1 Hour
  Cervical joint range of motion will be evaluated with a Universal goniometer. The pivot point will be placed on the C7 spinous process and the fixed arm will be kept perpendicular to the ground while the moving arm measures the movement of the cervical spinous process. The expected flexion angle is 45°.
Maximum Inspiratory Pressure Measurement | 1 Hour
  Measurements were taken with Pony Fx, mouth pressure measurement module Spirometer Device. After the appropriate filter and mouthpiece were attached to the spirometer, the nasal airway was closed with a clip. After inhaling against the completely closed airway for 20 seconds or for 10 breaths, the person was asked to inhale at the maximum rate at a time while sitting at the residual volume, to discharge the inhaled air from the nose. Measurement will be made again until the peak value is obtained., the highest value was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided